CLINICAL TRIAL: NCT06857695
Title: An Open-Label Study to Assess the Mass Balance Recovery, Absorption, Metabolism, Excretion of [14C]AZD5004 and Absolute Bioavailability of AZD5004 in Healthy Male Participants
Brief Title: A Study to Assess the Mass Balance and ADME of [14C]AZD5004 and the Absolute Bioavailability of AZD5004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7260C00010
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants
Keywords: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD5004 (Experimental): A single dose of AZD5004 film-coated tablet and a single dose of [14C]AZD5004 Solution for Infusion (Part 1)
  A single dose of [14C]AZD5004 Oral Solution (Part 2)
  Interventions: Drug: AZD5004 film-coated tablet; Drug: [14C]AZD5004 Solution for Infusion; Drug: [14C]AZD5004 Oral Solution

INTERVENTIONS:
Drug: AZD5004 film-coated tablet — oral, fasted
  Other Names: AZD5004
Drug: [14C]AZD5004 Solution for Infusion — intravenous, fasted
  Other Names: [14C]AZD5004
Drug: [14C]AZD5004 Oral Solution — oral, fasted
  Other Names: [14C]AZD5004

SUMMARY:
This study in healthy volunteers aims to answer these questions:

* Does the test medicine cause any important side effects?
* What are the blood levels of the test medicine and how quickly does the body get rid of it?
* How much of the test medicine taken by mouth gets into the bloodstream?
* How does the body break down and get rid of the test medicine?

This study will take place at one site in Nottingham, United Kingdom, and plans to enrol 8 healthy men aged 30-65 years, who will be involved in both parts of the study.

DETAILED DESCRIPTION:
In this 2-part study, healthy volunteers will be given three doses of test medicine to find out how the body breaks down and gets rid of the test medicine. Two doses will be 'radiolabelled' - they will contain a small amount of radioactivity (Carbon-14) so that it can be tracked in the body. The amount of radiactivity is less than 6 days of the average radiation exposure received in the UK each year, and slightly less than the radiation dose that would result from a single head x-ray or two leg x-rays.

This study in healthy volunteers aims to answer these questions:

* Does the test medicine cause any important side effects?
* What are the blood levels of the test medicine and how quickly does the body get rid of it?
* How much of the test medicine taken by mouth gets into the bloodstream?
* How does the body break down and get rid of the test medicine?

This study will take place at one site in Nottingham, United Kingdom.

It plans to enrol 8 healthy men aged 30-65 years, who will be involved in both parts of the study.

In Part 1, volunteers will receive a single dose of the test medicine by mouth and, on the same day, a very tiny dose of radiolabelled study medicine by injection into a vein. After a minimum of 7 days, in Part 2, volunteers will receive a dose of test medicine containing a very tiny amount of radio label, by mouth. They'll stay in the clinic for up to 6 nights in Part 1 and 8 nights in Part 2 and take up to 7 weeks to finish the study.

We'll collect blood and urine samples to do safety tests. Over a period of at least 15 days, we'll take many blood samples. In Part 2 volunteers will collect all their urine and faeces so that we can measure the amount of test medicine and its breakdown products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 30 to 65 years inclusive
* BMI in the range 18.0 - 35.0 kg/m2 and body weight ≥63 kg
* Regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History or presence of clinically significant gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity
* Excessive intake of caffeine containing drinks or food
* History/family history of medullary thyroid carcinoma or multiple endocrine neoplasia
* Uncontrolled thyroid disease
* History of acute pancreatitis or gallstones
* Serum triglyceride concentrations > 1000 mg/dL (11 mmol/L)
* Any history of significant inflammatory bowel disease, gastroparesis, or other severe disease or prior surgery affecting the upper GI tract
* Participants who do not have suitable veins for multiple venepunctures/cannulation
* Clinically significant abnormal clinical chemistry, haematology or urinalysis
* Significant hepatic disease
* Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG
* Abnormal renal function
* Radiation exposure exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years, occupationally exposed worker, or have been administered IMP in a [14C] ADME study in the last 12 months.
* Use of any prescribed or non-prescribed medication
* Current smokers or known or suspected history of alcohol or drug abuse.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability - Part 1 | Plasma sample collection from pre-dose to 110 hrs post-dose
  Absolute bioavailability (F) based on AUC0-inf of oral and IV administration, adjusted for dose
Amount of AZD5004 excreted (Ae) - Part 2 | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Mass balance recovery of total radioactivity (TR) in urine, faeces and all excreta (urine and faeces combined)
Amount of AZD5004 excreted expressed as a percentage of the dose administered (Fe) - Part 2 | Urine and faecal samples collected from pre-dose until 168 hours post dose
  Mass balance recovery of total radioactivity (TR) in urine, faeces and all excreta (urine and faeces combined)
Cumulative amount of AZD5004 excreted (CumAe) - Part 2 | Urine and faecal samples collected from pre-dose until 168 hours post dose
  Mass balance recovery of total radioactivity (TR) in urine, faeces and all excreta (urine and faeces combined)
Cumulative amount of AZD5004 excreted expressed as a percentage of the dose administered (CumFe) - Part 2 | Urine and faecal samples collected from pre-dose until 168 hours post dose
  Mass balance recovery of total radioactivity (TR) in urine, faeces and all excreta (urine and faeces combined)

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) for AZD5004 and total radioactivity (TR) - Part 1 and Part 2 | Plasma sample collection from pre-dose to 110 hours post-dose in Part 1 and from pre-dose to 168 hours post-dose in Part 2
  Pharmacokinetics (PK) ofAZD5004 and [14C]AZD5004 in plasma
Area under the curve from time 0 extrapolated to infinity (AUC0-inf) for AZD5004 - Part 1 and Part 2 | Plasma sample collection from pre-dose to 110 hours post-dose in Part 1 and from pre-dose to 168 hours post-dose in Part 2
  Pharmacokinetics (PK) of AZD5004 and [14C]AZD5004 in plasma
Area under the curve (AUC) of circulating plasma total radioactivity (TR) or accounting for 10% or more of the dose in excreta - Part 2 | Plasma, urine and faecal samples from pre-dose until 168 hours post-dose
  Identification of the chemical structure of each metabolite accounting for more than 10% by AUC of circulating total radioactivity (TR) or accounting for 10% or more of the dose in excreta
Blood:plasma concentration ratios - Part 2 | Whole blood and plasma samples collected from pre-dose until 168 hoours post-dose
  Blood:plasma concentration ratios for total radioactivity (TR)
Number of subjects with treatment-related adverse events - Part 1 and 2 | Through study duration, approximately 7 weeks
  To provide additional safety and tolerability information for AZD5004 by assessing the incidence of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual participant-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual participant-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/